CLINICAL TRIAL: NCT00736034
Title: A Single-Center, Open-Label Study to Assess the Efficacy of SharpPS™-Gold in Elderly Subjects With Memory Impairment
Brief Title: The Efficacy of Phosphatidylserine-Omega3 in Elderly Subjects With Memory Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Enzymotec (Industry)
Responsible Party: Inbal Eyal M.Sc, Enzymotec
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SharpPS™-Gold 001
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2010-03-24 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2009-04

CONDITIONS: Memory Impairment
Keywords: Age Associated Memory Impairment
MeSH Terms: conditions — Memory Disorders

INTERVENTIONS:
Dietary Supplement: Phosphatidylserine-Omega3 (SharpPS™-Gold) — Treatment will consist of capsules containing 100 mg phosphatidylserine-Omega3. Dosage: 1 capsule X 3 times daily, with meals. Duration: 15 weeks

SUMMARY:
The primary objective of this trial is to assess the ability of Phosphatidylserine-Omega3 to improve cognitive performance in elderly subjects with memory impairment.

This study is a single-center, open-label 15 weeks duration trial to assess efficacy of Phosphatidylserine-Omega3 in elderly subjects with memory impairment.

ELIGIBILITY:
INCLUSION CRITERIA

1. Ability to give written informed consent
2. Age: 90≥ years ≥65
3. Gender: male and female.
4. Clinical Dementia Rating Scale (CDR) ≤ 0.5
5. Mini-Mental State Examination (MMSE) ≥ 26
6. Memory test performance within or below the mean established for adults, with maximum of four neuropsychological subtests of the computerized test scored as 1.5 SD above the mean
7. Language: Subjects must be able to read, write and speak Hebrew.
8. Ability to perform tests and interviews.

EXCLUSION CRITERIA

1. Evidence of delirium, confusion, or other disturbances of consciousness.
2. Any Neurological disorder that could produce cognitive deterioration. Such disorders include AD, Parkinson's disease, stroke, intracranial hemorrhage, local brain lesions including tumors, and normal pressure hydrocephalus
3. History of any infective or inflammatory brain disease including those of viral, fungal, or syphilitic etiologies.
4. Head injury immediately preceding cognitive deterioration.
5. Current psychiatric diagnosis according to DSM IV criteria of depression, mania, or any other major psychiatric disorder, or evidence of depression as determined by the Geriatric Depression Scale (GDS15) score of 5 or more.
6. Current diagnosis or history of alcoholism or drug dependence.
7. Any medical disorder that could produce cognitive deterioration including renal, respiratory, cardiac and hepatic disease, diabetes mellitus, endocrine, metabolic or hematological disturbances unless well controlled, and malignancy not in remission for more than two years.
8. Use of psychotropic drug or any other drug or supplement that may significantly affect cognitive functioning during the month prior to psychometric testing.
9. Use of any experimental medication within 1 month prior to screening or as concomitant medications.
10. History of hypersensitivity or allergy to fish or fish oil.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Vakhapova, MD, Principal Investigator — Sourasky Medical Center
Locations (1):
- The Tel Aviv Sourasky Medical Center, Neurology department, Tel Aviv, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements in senior citizens' homes, hospitals, and newspapers.
Groups:
- PS-Omega3: Treatment will consist of capsules containing 100 mg phosphatidylserine-Omega3. Dosage: 1 capsule X 3 times daily, with meals
Period: Overall Study
Arm/Group | PS-Omega3
Started | 18
Completed | 16
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | PS-Omega3
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 75.29 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  Israel | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Neuropsychological Computerized Test
Description: The computerized neuropsychological assessment software consists of seven separate tasks: symbol spotting, pattern identification, pattern recall, digit-symbol substitution, digits span forward, digits span backward and delayed pattern recall. Based on the results obtained in the single tasks, eight cognitive composite scores are calculated including focused attention, sustained attention, memory recognition & recall, visuospatial learning, spatial short term memory, executive functions and mental flexibility.The total score range is from 0 to 100 points(0 is worse, 100 is best).
Time Frame: baseline, 15 weeks
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | PS-Omega3
Number analyzed (Participants) | 18
Points on a scale
  Focused Attention | 3.16 (12.39)
  Sustained Attention | -2.38 (11.09)
  Memory - Recognition | 1.88 (9.86)
  Memory - Recall | 4.50 (12.14)
  VisuoSpatial Learning | 8.83 (24.31)
  Spatial Short Term Memory | 13.16 (29.88)
  Executive Functions | -2.88 (19.72)
  Mental Flexibility | -3.88 (20.21)

2. Secondary Outcome: Clinical Global Impression of Change (CGI-C)Scale
Description: The Clinical Global Impression of Change (CGI-C)scale is designed to record the clinician's global impression of change. Global improvement score ranges from 1 = "Very much improved", through 4 = "No change", to 7 = "Very much worse". Participants who experienced an improvement (scores 1, 2 or 3) were classified as improved over the treatment period.
Time Frame: 15 weeks
Reporting Status: Not Posted
Measure: Number; unit: Participants who experienced improvement

ADVERSE EVENTS:
Arm/Group | PS-Omega3
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PS-Omega3 (N=18)
gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Hepatitis (General disorders) | 1 (1) — Not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No